CLINICAL TRIAL: NCT02297399
Title: Improvement of Tolerability for Bowel Preparation for Colonoscopy in Diabetic Patients. A Randomized Controlled Trial of Two Bowel Preparation Protocols Including 4 Liters PEG vs. 2 Liters PEG Plus Ascorbic Acid. iDIMEPREP Study.
Brief Title: Improvement of Tolerance of Bowel Cleansing Before Colonoscopy in Diabetic Patients
Acronym: iDIMEPREP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Marco Antonio Alvarez Gonzalez, MD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4790-I
Record Dates: First submitted 2014-11-13; First posted 2014-11-21 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus; Colonic Diseases
Keywords: Colonoscopy; Diabetes Mellitus; Polyethylene glycols; Ascorbate; Personal satisfaction
MeSH Terms: conditions — Diabetes Mellitus; Colonic Diseases; Personal Satisfaction | interventions — MoviPrep

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG-ascorbate 2L (Experimental): Subjects will take 2 liters of a polyethylene glycol 3500 (sodium sulphate, sodium chloride, postassium chloride), ascorbic acid and sodium ascorbate solution.
  Interventions: Drug: PEG-ascorbate 2L
- PEG 4L (Active Comparator): Subjects will take 4 liters of a polyethylene glycol 4000 (sodium sulphate, sodium chloride, postassium chloride and sodium bicarbonate) solution.
  Interventions: Drug: PEG 4L

INTERVENTIONS:
Drug: PEG-ascorbate 2L — Subjects will be asked to proceed to colonic cleansing with the interventional agents as per summary of product characteristics and specific instructions from members of the research team.
  Participants will be required to be on a low residue diet for 4 days before the procedure. The preparation will begin at 9:00 pm on the evening before the colonoscopy is scheduled. Participants will take 2 sachets (labelled A and B) of the investigational product and take their contents diluted in 1 liter of water. Two other sachets, also labelled A and B, will be taken diluted in 1 liter of water 4 to 5 hours before the procedure. Fasting will be required from 2 hours after the investigational product has been taken.
  Other Names: Moviprep®
  Arms: PEG-ascorbate 2L
Drug: PEG 4L — Subjects will be asked to proceed to colonic cleansing with the interventional agents as per summary of product characteristics and specific instructions from members of the research team.
  Participants will be required to be on a low residue diet for 4 days before the procedure. The preparation will begin at 9:00 pm on the evening before the colonoscopy is scheduled. Participants will take 8 sachets of the investigational product and take their contents diluted in 2 liters of water. Eight other sachets, also diluted in 2 liters of water will be taken 4 to 5 hours before the procedure. Fasting will be required from 2 hours after the investigational product has been taken.
  Other Names: Bohm®
  Arms: PEG 4L

SUMMARY:
This trial will compare the tolerance to 2 different methods for colon cleansing before colonoscopy in diabetic patients.

DETAILED DESCRIPTION:
Consecutive diabetic patients undergoing an ambulatory colonoscopy at the participating sites will be randomized to 2 different methods of colon cleansing before the procedure.

Both will be based on the oral ingestion of a fluid solution (half of it on the evening before the procedure is planned and the rest on the morning of the same day), and the main difference between them will be the volume of fluid that will be ingested in each case.

Analogic visual scales and standardized questionnaires on various aspects that may influence the degree of satisfaction about the preparation will be answered by the participants and collected before the colonoscopy. The endoscopist, blinded to the preparation method, will grade the adequacy of the preparation. Adverse events will be recorded up to 1 month after the procedure

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a diagnostic, screening or follow-up outpatient colonoscopy
* Diabetes mellitus (being treated with insulin or any oral agent).

Exclusion Criteria:

* Unwillingness to participate.
* Hospital admission at the time of colonoscopy.
* Inability to follow instructions
* Active inflammatory bowel disease
* Previous colectomy.
* Incomplete colonoscopies due to technical reasons or contraindication for the procedure as evaluated by the endoscopist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2016-01-26 (Actual); Study Completion 2016-01-26 (Actual)

PRIMARY OUTCOMES:
Tolerability of the bowel preparation (analogue visual scale) | 6 hours after finishing bowel preparation
  Each participant will rate his/her experience in an analogue visual scale.

SECONDARY OUTCOMES:
Ease of consumption and taste of the laxative (analogue visual scale) | 6 hours after finishing bowel preparation
  Each participant will rate his/her experience in an analogue visual scale.
Abdominal pain, nausea and bloating (analogue visual scale) | 6 hours after finishing bowel preparation
  Each participant will rate his/her experience in an analogue visual scale.
Acceptability of the preparation (interference with work, leisure activities or sleep questionnaire) | 6 hours after finishing bowel preparation
  Each participant will rate his/her experience in a questionnaire.
Adherence to the planned bowel cleansing method (questionnaire) | 6 hours after finishing bowel preparation
  Each participant will rate his/her experience in a questionnaire.
Efficacy of the bowel preparation (Boston Bowel Preparation Scale (BBPS) | 10 minutes after the colonoscopy
  Rating of the Boston Bowel Preparation Scale (BBPS) by the endoscopist
Adverse events | 30 days after the colonoscopy
  Description of any adverse event occurred during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Marco Antonio Alvarez González, MD, PhD, Principal Investigator — Parc de Salut Mar
Locations (2):
- Spain (2):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona

REFERENCES:
- [Background] Hsu CW, Imperiale TF. Meta-analysis and cost comparison of polyethylene glycol lavage versus sodium phosphate for colonoscopy preparation. Gastrointest Endosc. 1998 Sep;48(3):276-82. doi: 10.1016/s0016-5107(98)70191-9. PMID 9744604
- [Background] Aronchick CA, Lipshutz WH, Wright SH, Dufrayne F, Bergman G. A novel tableted purgative for colonoscopic preparation: efficacy and safety comparisons with Colyte and Fleet Phospho-Soda. Gastrointest Endosc. 2000 Sep;52(3):346-52. doi: 10.1067/mge.2000.108480. PMID 10968848
- [Background] Taylor C, Schubert ML. Decreased efficacy of polyethylene glycol lavage solution (golytely) in the preparation of diabetic patients for outpatient colonoscopy: a prospective and blinded study. Am J Gastroenterol. 2001 Mar;96(3):710-4. doi: 10.1111/j.1572-0241.2001.03610.x. PMID 11280539
- [Background] Ozturk NA, Gokturk HS, Demir M, Erdogan D, Unler GK, Gur G, Yilmaz U. The effect of autonomous neuropathy on bowel preparation in type 2 diabetes mellitus. Int J Colorectal Dis. 2009 Dec;24(12):1407-12. doi: 10.1007/s00384-009-0757-4. Epub 2009 Jul 7. PMID 19582466
- [Background] Ell C, Fischbach W, Bronisch HJ, Dertinger S, Layer P, Runzi M, Schneider T, Kachel G, Gruger J, Kollinger M, Nagell W, Goerg KJ, Wanitschke R, Gruss HJ. Randomized trial of low-volume PEG solution versus standard PEG + electrolytes for bowel cleansing before colonoscopy. Am J Gastroenterol. 2008 Apr;103(4):883-93. doi: 10.1111/j.1572-0241.2007.01708.x. Epub 2008 Jan 11. PMID 18190651